CLINICAL TRIAL: NCT06172257
Title: A Phase 3 Double-masked, Randomized, Multicenter Study of the Efficacy and Safety of OCS 01 Eye Drops in Subjects With Diabetic Macular Edema
Brief Title: A Pivotal Safety and Efficacy Study of OCS-01 Eye Drops in Participants With Diabetic Macular Edema (DIAMOND 2)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oculis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DX221
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Macular Edema
Keywords: Topical ophthalmic suspension; Eye drop
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OCS-01 (Experimental): dexamethasone ophthalmic suspension,1.5% [15 mg/mL]
  Interventions: Drug: Dexamethasone ophthalmic suspension (OCS-01)
- Vehicle ophthalmic suspension (Placebo Comparator): Vehicle of OCS-01
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Dexamethasone ophthalmic suspension (OCS-01) — Participants will be dosed with one eye drop of OCS-01 6 times per day for 6 weeks (induction phase) followed by 3 times per day for 46 weeks (maintenance phase).
  Other Names: Dexamethasone
  Arms: OCS-01
Drug: Vehicle — Participants will be dosed with one eye drop of vehicle 6 times per day for 6 weeks (induction phase) followed by 3 times per day for 46 weeks (maintenance phase).
  Other Names: Placebo
  Arms: Vehicle ophthalmic suspension

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of the topical ophthalmic administration of OCS 01 as compared to Vehicle in participants with Diabetic Macular Edema (DME).

DETAILED DESCRIPTION:
A Phase 3 Pivotal Double-masked, Randomized, Vehicle-controlled, Multicenter Study of the Efficacy and Safety of OCS 01 Eye Drops in participants with Diabetic Macular Edema

ELIGIBILITY:
Inclusion Criteria (selection):

1. Have a signed informed consent form before any study-specific procedures are performed.
2. Have DME with presence of intraretinal and/or subretinal fluid in the study eye, with CST of ≥310 µm by SD-OCT at screening (Visit 1) (as assessed by an independent reading center).
3. Have a documented diagnosis of Type 1 or Type 2 diabetes mellitus prior to screening (Visit 1).

Exclusion Criteria (selection):

1. Have macular edema considered to be because of a cause other than DME.
2. Have a decrease in BCVA because of causes other than DME.
3. Have a known history of significant macular ischemia which would prevent gain in visual acuity in the study eye.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in BCVA (Best Corrected Visual Acuity) | Week 52
  Assessed using ETDRS (Early Treatment Diabetes Retinopathy Study) letters score: higher numbers on the ETDRS chart representing better visual acuity.

SECONDARY OUTCOMES:
Percentage of Participants With a 3-line or Greater Gain in BCVA | Baseline, Week 52
  BCVA will be assessed using ETDRS letters score: higher numbers on the ETDRS chart representing better visual acuity.
Mean Change in BCVA | Baseline, Week 12 and Week 24
  BCVA will be assessed using ETDRS letters score: higher numbers on the ETDRS chart representing better visual acuity.
Mean Change in Central Subfield Thickness (CST) | Baseline, Week 52
  CST will be measured by spectral domain optical coherence tomography (SD-OCT)

OTHER OUTCOMES:
Number of Participants with Treatment Emergent Adverse events (TEAEs) | Up to Week 52
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant. TEAEs are those AEs that occur after administration of the study product and are therefore temporally associated with the use of the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Do, MD, Principal Investigator — Stanford Byers Eye Institute
Locations (62):
- United States (42):
  - Associated Retina Consultants, Gilbert, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Consultants of Arizona - Phoenix North, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina Associates of Southern California, Huntington Beach, California
  - Stanford Byers Eye Institute, Palo Alto, California
  - Retinal Consultants Medical Group, Inc, Sacramento, California
  - Retinal Consultants Medical Group, Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - Macula Retina Vitreous Center, Torrance, California
  - Retina Specialists of Colorado, Denver, Colorado
  - Eye Care Center of Northern Colorado, Longmont, Colorado
  - Sibia Eye Institute, Boynton Beach, Florida
  - Blue Ocean Clinical Research, Clearwater, Florida
  - Advanced Research, Coral Springs, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Retina Consultants of Southwest Florida, Naples, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - Georgia Retina, Peachtree City, Georgia
  - Illinois Retina Associates, Oak Park, Illinois
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Mississippi Retina Associates, Jackson, Mississippi
  - Sierra Eye Associates, Reno, Nevada
  - VitreoRetinal Consultants of NY, Hauppauge, New York
  - Island Retina, Shirley, New York
  - Vitreoretinal Consultants of NY, Westbury, New York
  - Erie Retina Research, Erie, Pennsylvania
  - Vision Research Solutions in Philadelphia, Philadelphia, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina, Nashville, Tennessee
  - Retina Consultants of Texas, Bellaire, Texas
  - Star Retina, Burleson, Texas
  - Houston Eye Associates, North Loop, Houston, Texas
  - Austin Retina Associates, Round Rock, Texas
  - San Antonio Eye Center - Downtown Clinic, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Tyler Retina Consultants, Tyler, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
- Argentina (13):
  - Fundacion Zambrano, Buenos Aires, Buenos Aires
  - Oftalmos - Instituto Oftalmológico de Alta Complejidad, Buenos Aires, Buenos Aires
  - Centro De Ojos Loria Srl, CABA, Buenos Aires
  - Centro Privado de Ojos, CABA, Buenos Aires
  - Organizacion Medica De Investigacion, CABA, Buenos Aires
  - Buenos Aires Macula (BAM) Clinical Research, CABA, Buenos Aires
  - Charles Centro Oftalmológico, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Centro Privado de Ojos Romagosa, Córdoba, Córdoba Province
  - Instituto de Microcirugía Ocular Córdoba (IMOC), Córdoba, Córdoba Province
  - Oftar Mendoza - Centro Privado de Oftalmología en Mendoza Capital, Mendoza, Mendoza Province
  - Centro de la Vision Dr. Kolton, Salta, Salta Province
  - Grupo Laser Vision, Rosario, Santa Fe Province
  - Oftalmologìa Global, Rosario, Santa Fe Province
- India (6):
  - Rising Retina Clinic, Ahmedabad, Gujarat
  - Narayana Nethralaya, Bangalore, Karnataka
  - Agrawal Hospital, Jaipur, Rajasthan
  - Lotus Eye Hospital and Institute, Coimbatore, Tamil Nadu
  - St. Theresa's Hospital, Hyderabad, Telangana
  - GSVM Medical College, Kanpur, Uttar Pradesh
- Emanuelli Research & Development Center, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No